CLINICAL TRIAL: NCT04303897
Title: A Real-World Evidence Study to Evaluate the Safety and Effectiveness of XEN Glaucoma Treatment System (XEN) in Chinese Patients With Refractory Glaucoma
Brief Title: Real-world Evidence Study of XEN in Chinese Patients With Refractory Glaucoma
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 1924-801-007
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Refractory Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- XEN Glaucoma Stent
  Interventions: Device: XEN Glaucoma Stent

INTERVENTIONS:
Device: XEN Glaucoma Stent — Data are collected from patients who are implanted with XEN via the specific urgent medical needs for named patient use regulatory pathway in Hainan

SUMMARY:
Real-world evidence study to assess the safety and effectiveness of XEN® Glaucoma Treatment System in Chinese patients with refractory glaucoma. Participants will be (prospective) or have already been (retrospective) implanted with XEN via specific urgent medical need.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory glaucomas, including cases where previous surgical treatment has failed, cases of POAG, and pseudoexfoliative or pigmentary glaucoma with open angles that are unresponsive to maximum tolerated medical therapy

Exclusion Criteria:

* Angle closure glaucoma where angle has not been surgically opened
* Previous glaucoma shunt/valve in the target quadrant
* Presence of conjunctival scarring, prior conjunctival surgery or other conjunctival pathologies (eg, pterygium) in the target quadrant
* Active inflammation (eg, blepharitis, conjunctivitis, keratitis, uveitis)
* Active iris neovascularization or neovascularization of the iris within six months of the surgical date
* Anterior chamber intraocular lens
* Presence of intraocular silicone oil
* Vitreous present in the anterior chamber

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are being implanted with the approved XEN product via the specific urgent medical needs for named patient use regulatory pathway in Hainan. The XEN Glaucoma Treatment System (XEN) is comprised of the XEN45 Gel Stent and XEN® Injector.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving at least a 20% reduction from intraocular pressure (IOP) while on the same number or fewer number of IOP lowering medications than at baseline | Baseline to Month 12

SECONDARY OUTCOMES:
Mean decrease in IOP | Baseline to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (1):
- Boao Super Hospital /ID# 233669, Qionghai, Hainan, China

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=1924-801-007#additional-resources-section